CLINICAL TRIAL: NCT06821230
Title: Enhancing Psychological Wellbeing and the Patient-caregiver Relationship Through Dyadic Mindfulness: a Randomized Controlled Trial in People with Parkinson's Disease and Their Caregivers
Brief Title: Dyadic Mindfulness for People with Parkinson's Disease and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok Yan Yan, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 17605424
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Mindfulness; Caregivers; Movement Disorders; Neurodegenerative Disease; Dyadic Intervention; Psychosocial Health; Parkinsons Disease
Keywords: Parkinsons disease; Mindfulness; dyadic care
MeSH Terms: conditions — Movement Disorders; Neurodegenerative Diseases; Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dyadic mindfulness group (Experimental)
  Interventions: Behavioral: Dyadic mindfulness
- Wait-list usual care control group (No Intervention): The wait-list, usual care control group will continue with routine outpatient services (medication follow-up care with minimal health education on disease management/drug care) and then receive dyadic mindfulness training after the 6-month study period.

INTERVENTIONS:
Behavioral: Dyadic mindfulness — The dyadic mindfulness intervention group will receive 8 weekly 90-min sessions, with a total of 12 contact hours. The intervention will be delivered in a small group format with 6-8 dyads each and led by a certified yoga instructor with mindfulness qualifications. The program content mindfulness meditation, mindful breathing, and yoga sequences with warm-up and cool-down and each component is modified to pair-based practices.
  Arms: Dyadic mindfulness group

SUMMARY:
The proposed two-arm randomized waitlist-controlled trial will use a mixed-methods design to investigate the effects of dyadic mindfulness on physio-psycho-spiritual outcomes in people with Parkinson's Disease (PwPD) and their family caregivers. One hundred Chinese patient-caregiver dyads will be randomized to receive eight weekly 90-minute dyadic mindfulness sessions or usual care. Outcome measures include negative emotions (primary outcome), patient-caregiver relationship, mindfulness, HRQOL, gut microbiome, PD-related symptoms, and caregiving burden. An actor-partner interdependence model will be used to explore the interactions of treatment effects within the dyads. The dyads will be assessed at baseline(T0), post-intervention(T1), and 4-months post-intervention(T2). The investigators will also invite 25 dyads to attend in-depth interviews exploring their experiences, perceived changes, and factors attributable to the effectiveness/ineffectiveness of the intervention. Generalized linear mixed-effects (GLME) with intention-to-treat analysis will be used to compare the changes in outcomes over time within and between the two arms. The findings will be triangulated to provide a comprehensive evaluation of the intervention's effectiveness. This study will generate rigorous scientific evidence to inform the application of dyadic mindfulness as a public health practice preventing the progression of psychological distress in PwPD and caregivers to clinically severe levels. Its self-help nature also enriches the primary care for this clinical cohort.

ELIGIBILITY:
Inclusion Criteria of PwPD:

* Chinese patients with idiopathic mild-moderate PD (as indicated by the Hoehn and Yahr Scale stages I-III: those with unilateral/bilateral symptoms, with/without postural instability who are able to walk/stand unassisted)
* Aged 50-80
* Experience at least mild negative emotions (as indicated by the 21-item Depression, Anxiety and Stress Scale [DASS21] score of Depression subscale ≥10, Anxiety subscale ≥8, or Stress subscale ≥15)

Inclusion Criteria of caregivers of PwPD:

- Self-identified as the primary caregivers of their patient

Both need to be able to communicate in Cantonese and provide written consent.

Exclusion Criteria:

* Engage in regular supervised mind-body practices such as Tai Chi, yoga, or other forms of mindfulness training (>2 times per week)
* Have a pre-existing acute psychotic disease
* Currently participating in any other behavioral or pharmacological trial
* Have significant cognitive impairment, as indicated by an Abbreviated Mental Test score≤ 6
* Have other contraindications that may limit their full participation (e.g., severe hearing/vision impairment)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Negative emotions | A repeated outcome measure will be conducted at baseline (T0, prior to randomization), immediate post-intervention (T1, 2 months) and 4-months post-intervention (T2, 6 months).
  Negative emotions (primary outcome) will be measured by validated Chinese DASS-21 using a one-week recall period, which was developed to measure three related and clinically significant negative emotional states of depression, anxiety and stress. Each item is rated on a 0-3 scale (0="Did not apply to me at all" to 3="Applied to me very much or most of the time"). The score of each subscale ranges from 0-42 and the total score ranges from 0-126, with higher score indicating greater self-reported levels of depression, anxiety and stress.

SECONDARY OUTCOMES:
Patient-caregiver relationship | A repeated outcome measure will be conducted at baseline (T0, prior to randomization), immediate post-intervention (T1, 2 months) and 4-months post-intervention (T2, 6 months).
  Patient-caregiver relationship will be measured by the validated Chinese Dyadic Relationship Scale, which comprises two subscales: dyadic strain and positive dyadic interaction. Each item is rated on a four-point Likert-type scale ranging from 0 (strongly agree) to 3 (strongly disagree).
Mindfulness | A repeated outcome measure will be conducted at baseline (T0, prior to randomization), immediate post-intervention (T1, 2 months) and 4-months post-intervention (T2, 6 months).
  Mindfulness will be measured by the validated Chinese 32-item Multidimensional Assessment of Interoceptive Awareness (MAIA). 36 Using a six-point Likert scale, eight domains will be assessed: noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening and trusting.
HRQOL | A repeated outcome measure will be conducted at baseline (T0, prior to randomization), immediate post-intervention (T1, 2 months) and 4-months post-intervention (T2, 6 months).
  HRQOL will be measured by the validated Chinese EuroQol 5-dimension 5-level questionnaire (EQ-5D-5L). It comprises 2 main components: a description of health status in 5 dimensions (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression), and a numeric value of overall health status perceived by the respondents (EQ-VAS). Each dimension is scored on a 5-point Likert scale, from 0 (no problems) to 4 (extreme problems). The EQ-VAS records an individual's self-rated health on a numeric analogue visual scale from 0 (the worst health) to 100 (the best health).
Gut microbiome | A repeated outcome measure will be conducted at baseline (T0, prior to randomization), immediate post-intervention (T1, 2 months) and 4-months post-intervention (T2, 6 months).
  Gut microbiome. All participants will be instructed to self-collect a fecal sample any time during the week of the study visits. Samples will be kept in a collection tube with a stabilizer and stored at room temperature. The fecal sample collection procedure will be guided by a previously tested information leaflet and YouTube video. The research team will collect the samples during the study visits and transfer them to labeled cryovials within 60 days of collection according to the manufacturer's protocol. The samples will then be stored at -80◦C until further analysis.
PD-related motor and non-motor symptoms | A repeated outcome measure will be conducted at baseline (T0, prior to randomization), immediate post-intervention (T1, 2 months) and 4-months post-intervention (T2, 6 months).
  PD-related motor and non-motor symptoms will be measured by the validated Movement Disorder Society-Unified Parkinson's Disease Rating Scale (Chinese) Parts I-III, which examine non-motor experiences, motor experiences of daily living, and clinical examination of motor symptoms, respectively. Higher scores indicate greater disease severity.
Caregiving burden | A repeated outcome measure will be conducted at baseline (T0, prior to randomization), immediate post-intervention (T1, 2 months) and 4-months post-intervention (T2, 6 months).
  Caregiving burden will be made using the validated 12-item Zarit Burden Interview-short version, which assesses three domains on a five-point scale (0= "never"; 4="very frequently"): perceived role strain, self-criticism, and negative emotion. Higher scores indicate a heavier caregiving burden.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data supporting the findings of this study are available upon request from the principal investigator, Prof. Kwok. These data are not publicly available, as they contain information that could compromise the privacy of research participants.